CLINICAL TRIAL: NCT03747978
Title: Short-term Effects of Perindopril-amlodipine Versus Perindopril-indapamide on Blood Pressure Control in Newly Diagnosed Type 2 Diabetes Individuals With Hypertension
Brief Title: Short-term Effects of Perindopril-amlodipine Versus Perindopril-indapamide in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, Sobngwi Eugene, Medical Advisor, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNO20164
Record Dates: First submitted 2018-11-18; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: diabetes; hypertension; blacks; Africa; ACE inhibitor; Calcium channel blocker; Diuretic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus | interventions — amlodipine, perindopril drug combination; indapamide, perindopril drug combination

STUDY DESIGN:
Intervention Model Description: double blind head to head trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perindopril and Amlodipine (Experimental): Fixed dose combination of Perindopril 5mg and Amlodipine 5mg tablets once daily for 6 weeks
  Interventions: Drug: Perindopril and Amlodipine
- Perindopril-Indapamide (Active Comparator): Fixed-dose combination of Perindopril 5mg and Indapamide 1.25mg tablets once daily for 6 weeks
  Interventions: Drug: Perindopril-indapamide

INTERVENTIONS:
Drug: Perindopril and Amlodipine — Fixed combination of Perindopril 5mg and Amlodipine 5mg
  Other Names: Coveram5/5mg
  Arms: Perindopril and Amlodipine
Drug: Perindopril-indapamide — Perindopril 5mg and Indapamide 1.25mg
  Other Names: Bipreterax5/1.25
  Arms: Perindopril-Indapamide

SUMMARY:
This was a double-blinded randomized controlled trial of 24-hour blood pressure control in sub Saharan type 2 diabetes patients, newly diagnosed for hypertension. They were allocated to receive either a fixed combination of perindopril + amlodipine or perindopril + indapamide for 42 days.

DETAILED DESCRIPTION:
This was a double-blinded randomized controlled trial conducted at the National Obesity Center and the cardiology unit of the Yaoundé Central Hospital in Cameroon from October 2016 to May 2017. Eligible patients were type 2 diabetes patients, newly diagnosed for hypertension (grade I or II) with confirmation on ambulatory BP monitoring (ABPM). Patients were either on lifestyle modification alone or on a stable anti-diabetic treatment for the past three months, aged 25-65 years naïve to any anti-hypertensive treatment, who provided their written informed consent. Participants were assigned to receive as anti-hypertensive treatment perindopril-amlodipine once daily or perindopril-indapamide at the same frequency. The two groups were followed up and monitored for sixth weeks and patients did not take any additional treatment with BP modifying properties.

The primary outcome was the relative change in circadian blood pressure profile between the two groups after six weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* adult diabetes patients aged between 25-65 years,
* with grade I or grade II (WHO classification) hypertension on the clinical measure, confirmed by ABPM
* naïve to any anti-hypertensive treatment
* written informed consent.

Exclusion Criteria:

* Patients with grade III hypertension (WHO classification) were classified as hypertensive emergency,
* estimated creatinine clearance ˂30ml/min/1.73m2 (using Modified Diet in Renal Diseases formula)
* alanine transaminase (ALT)≥ 3 normal
* any contraindication to study drugs (hypersensitivity)
* pregnant or breastfeeding women

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
24-hour blood pressure | 6 weeks
  Change in average 24-hour blood pressure

SECONDARY OUTCOMES:
night blood pressure dip | 6 weeks
  Change in average night time blood pressure drop

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sobngwi, MD, PhD, Principal Investigator — Yaounde Central Hospital
Locations (1):
- National Obesity Centre, Yaounde Central Hospital, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sobngwi E, Mfeukeu-Kuate L, Kouam M, Tankeu AT, Nganou-Gnindjio CN, Hamadou B, Etoa M, Ngassam E, Nkamgna A, Dehayem MY, Kaze FF, Kengne AP, Mbanya JC. Short-term effects of perindopril-amlodipine vs perindopril-indapamide on blood pressure control in sub-Saharan type 2 diabetic individuals newly diagnosed for hypertension: A double-blinded randomized controlled trial. J Clin Hypertens (Greenwich). 2019 Jul;21(7):1002-1008. doi: 10.1111/jch.13557. Epub 2019 Jun 8. PMID 31175711